CLINICAL TRIAL: NCT03830580
Title: Benefit of Singing in the Care of Premature Children Undergoing Screening for Retinopathy of Prematurity in the Neonatology and Neonatal Resuscitation Unit of the Dijon University Hospital
Acronym: Voix Chantée
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHARY-TARDY 2018
Record Dates: First submitted 2019-01-25; First posted 2019-02-05 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Prematurity; Eye Fundus
MeSH Terms: conditions — Premature Birth | interventions — Singing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sung voice (Experimental)
  Interventions: Other: Positive stimulation (singing)
- Control (No Intervention)

INTERVENTIONS:
Other: Positive stimulation (singing) — A nurse or assistant trained in singing with an operal singer sings a lullaby She sits next to the incubator and sings from the time the sucrose is administered (2 minutes before the fundus exams is performed) until the end of the examination - taking into account the child's reaction
  Arms: Sung voice

SUMMARY:
As part of the regular procedure for premature births, premature infants undergo several screening examinations, including an examination of the fundus. This examination seeks to establish whether the infant has retinopathy of prematurity. This disease affects the vessels of the retina of the eye, especially in prematurely born children, and can lead to serious complications such as blindness if it is not treated in time.

The purpose of this study is to assess the discomfort caused by the screening in order to improve practices. To do this, the investigators would like to evaluate whether soft auditory stimulation, more precisely a person singing, would improve the children's level of comfort during the examination.

To do this, the participating children will be divided into 2 groups:

* The "Singing" group will receive the usual comfort treatments (placed in a 'nest', pacifier and sugar water) and a trained professional will sing a lullaby or nursery rhyme at the same time
* control group will receive the usual comfort care (placed in a 'nest', pacifier and sugar water) The child's head and entire body will be filmed, which will allow an evaluator to assess the child's comfort.

ELIGIBILITY:
Inclusion Criteria:

* Infant born prematurely before the end of 31 weeks of amenorrhoea and/or with a birth weight of less than 1250g
* Infant in whom a first screening examination (fundus) for retinopathy of prematurity (i.e. around 32 WA) must be carried out according to term by hospital protocol
* Infant hospitalized in the neonatal paediatrics and intensive care unit of the Dijon University Hospital
* Infant affiliated to the national medical insurance system
* Oral agreement of one of the two parents

Exclusion Criteria:

* Infants with contraindications to the use of Algopedol® 24% sugar solution, NEOSYNEPHRINE 2.5% mydriatic eye drops for pupillary dilatation, MYDRIATICUM 0.5% mydriatic eye drops for pupillary dilatation and OXYBUPROCAINE analgesic eye drops
* Infant with known deafness and no hearing aid
* Premature infant in critical condition
* Infant with hemodynamic and clinical instability making it impossible to perform the fundus examination because of the risk of decompensation
* Parent refuses the videotaping

Ages: 1 Month to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Acute pain assessed by the PIPP (Premature Infant Pain Profile) scale | During the examination
  The children's faces and bodies will be filmed - without sound - during the examination. The nurse who examines the fundus will start and finish the video recording.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France